CLINICAL TRIAL: NCT00970242
Title: Ambulatory Urodynamic Evaluation of Sacral Neuromodulation for Non-obstructive Urinary Retention
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sajjad Rahnama'i, department of Urology
Other Study IDs: MEC 09-4-053
Record Dates: First submitted 2009-09-01; First posted 2009-09-02 (Estimated); Last update posted 2009-09-04 (Estimated); Status verified 2009-09

CONDITIONS: Acontractile Bladder

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Ambulatory Urodynamic measurement on patients with diminished or absent bladder contractility before and after trial with Sacral Neuromodulation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diminished or absent bladder contraction

Exclusion Criteria:

* Prior Neuromodulation therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with diminished or absent bladder contraction
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2009-08; Primary Completion 2012-01 (Estimated); Study Completion 2012-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Sajjad Rahnama'i, MD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- MaastrichtUMC, Maastricht, Netherlands